CLINICAL TRIAL: NCT00779324
Title: A Multi-Center, Parallel-Group, Randomized, Double-Blind, Placebo-Controlled Trial of Amantadine Hydrochloride in the Treatment of Chronic Traumatic Brain Injury Irritability and Aggression: A Replication Study
Brief Title: Amantadine for the Treatment of Traumatic Brain Injury Irritability and Aggression: A Multi-site Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Indiana University (Other); University of Washington (Other); The Institute for Rehabilitaion and Research Foundation (Other); Spaulding Rehabilitation Hospital (Other); Ohio State University (Other); Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 09-08-11B; H133A080035 (Other Grant/Funding Number: NIDRR)
Record Dates: First submitted 2008-10-23; First posted 2008-10-24 (Estimated); Results first posted 2021-09-10 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2021-08

CONDITIONS: Brain Injury; Aggression
Keywords: traumatic brain injury; irritability; aggression; amantadine; behavior
MeSH Terms: conditions — Brain Injuries; Aggression; Brain Injuries, Traumatic; Behavior | interventions — Amantadine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Amantadine (Experimental): Amantadine 100 mg every morning and Noon
  Interventions: Drug: Amantadine Hydrochloride
- Placebo (Placebo Comparator): Placebo tablets
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Amantadine Hydrochloride — 100 mg every morning and noon
  Other Names: Symmetrel
  Arms: Amantadine
Drug: Placebo — one placebo tablet every morning and 12 Noon
  Arms: Placebo

SUMMARY:
The purpose of this study is to study the effect of amantadine on irritability and aggression caused by traumatic brain injury.

DETAILED DESCRIPTION:
PURPOSE OF PROJECT: To study the effect of amantadine 100 mg administered twice daily compared to placebo on irritability from baseline to treatment Day 28.

SUMMARY OF PROJECT: It is anticipated that 168 subjects with 168 corresponding subject informants will be recruited for the study. Carolinas Rehabilitation, the lead center, and 5 collaborating centers will enroll approximately 28 subjects each.

Subjects will be recruited primarily from the clinics. Also, letters will be sent to patients in our data base. If the first encounter with research personnel is by telephone, the research assistant will obtain verbal (telephone) consent from the subject's informant for the Neuropsychiatric Inventory (NPI) for subject irritability. The score on this questionnaire must be ≥ 6 for qualification. This allows pre-screening to take place and avoid an unnecessary clinic visit.

Subjects who consent and qualify will be randomized in a 1:1 ratio, amantadine to placebo. Stratification to randomization group will occur based on the presence of depression defined by a Beck's Depression Inventory-II (BDI-II) score ≥ 13. Randomized subjects will receive amantadine or placebo 100 mg twice daily every morning and 12 Noon. There will be 4 clinic visits. Visits will occur at baseline, for consenting and screening, day 28, day 60 and day 90. At all 4 clinic visits, both the subject and the informant will be given questionnaires regarding the subject's behavior and mood. Follow up phone calls will occur each week that the subject is not seen in the clinic until the end of the study. Follow up phone calls will assess for study medication compliance, adverse events and concomitant medication changes. Day 60 ends the period of the Randomized Clinical Trial phase of the study and the subjects will begin the 1 month continuation phase of the study when all participants receive active amantadine.

The following questionnaires will be used as measures of irritability for the subject and the informant: Neuropsychiatric Inventory (NPI), State Trait Anger Expression Inventory (STAXI-2), and Global Impression of Change.

The following questionnaires will be dispensed to the subject only: Short Form -12, Satisfaction With Life Scale, Patient Health Questionnaire, Beck Depression Inventory, Brief Symptom Inventory, Family Assessment Device, Fatigue Impact Scale, and tests of cognitive function. The Glasgow Outcome Score-Extended will be completed by the research assistant using information obtained primarily from the informant.

The Investigator will complete the Clinical Global Impression of change at Visits 1, 2, 3, and 4.

History and Physical Exam, creatinine level (kidney function) will be obtained for safety and tolerability. Serum pregnancy tests will be drawn at screening for females of childbearing potential.

ELIGIBILITY:
Inclusion Criteria:

* Closed head injury (defined as impaired brain function resulting from externally inflicted trauma without penetrating injury) at least 6 months prior to enrollment
* Irritability that is either new or worse than the level of irritability before the traumatic brain injury, by report of the Observer or person with TBI
* Age at time of enrollment: 16 to 75 years
* Voluntary informed consent and authorization of participant and informant
* Subject and informant willing to comply with the protocol
* Informant-rated NPI Irritability Domain score 6 or greater (moderate-to-severe irritability)
* Medically and neurologically stable during the month prior to enrollment
* If taking antidepressant, anxiolytic, hypnotic, or stimulant medications, no change anticipated in these medications during the month prior to enrollment or during the 90-day participation
* No change in therapies or medications planned during the 90-day participation
* No surgeries planned during the 90-day participation
* Vision, hearing, speech, motor function, and comprehension sufficient to complete interviews
* Observer (e.g.: family member, close friend, employer) with whom subject interacts sufficiently to observe occurrences of irritability. The observer interacts with the participant for a period long enough and of a nature to be able to judge the participant's irritability. The interactions would need to be adequate to judge observer distress over the irritability, severity of irritability and frequency of irritability on the following scale: < once weekly; once per week; several times per week, but not every day; essentially continuous.

Exclusion Criteria:

* Previous participation in the Carolinas TBI Model System amantadine irritability study
* Ingestion of amantadine hydrochloride during the month prior to enrollment
* Potential subject without a reliable informant
* Penetrating head injury as defined by head injury due to gunshot, projectile or foreign object
* Injury < 6 months prior to enrollment
* Inability to interact sufficiently for communication with caregiver
* Clinical signs of active infection
* Diagnosis of seizure in the month prior to enrollment
* Creatinine clearance <60 mL/min
* Pregnancy (Beta-HCG + females of child-bearing potential) and lactating females
* Concurrent use of first generation neuroleptic agents or phenelzine
* History of schizophrenia or psychosis
* Active concern of schizophrenia or psychosis
* Diagnosis of progressive or additional neurologic disease that affects brain function, except stroke that occurs at th same time as the TBI
* Previous allergy or adverse reaction to amantadine hydrochloride

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2009-08; Primary Completion 2013-04 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Flora M Hammond, MD, Principal Investigator — Carolinas Rehabilitation
Locations (6):
- United States (6):
  - Indiana University and the Rehabilitation Hospital of Indiana, Indianapolis, Indiana
  - Spaulding Rehabilitation, Boston, Massachusetts
  - Carolinas Rehabilitation, Charlotte, North Carolina
  - The Ohio State University, Columbus, Ohio
  - TIRR Memorial Herman, Houston, Texas
  - University of Washington, Seattle, Washington

REFERENCES:
- [Derived] Hammond FM, Sherer M, Malec JF, Zafonte RD, Dikmen S, Bogner J, Bell KR, Barber J, Temkin N. Amantadine Did Not Positively Impact Cognition in Chronic Traumatic Brain Injury: A Multi-Site, Randomized, Controlled Trial. J Neurotrauma. 2018 Oct 1;35(19):2298-2305. doi: 10.1089/neu.2018.5767. Epub 2018 Jun 7. PMID 29742960
- [Derived] Hammond FM, Malec JF, Zafonte RD, Sherer M, Bogner J, Dikmen S, Whitney MP, Bell KR, Perkins SM, Moser EA. Potential Impact of Amantadine on Aggression in Chronic Traumatic Brain Injury. J Head Trauma Rehabil. 2017 Sep/Oct;32(5):308-318. doi: 10.1097/HTR.0000000000000342. PMID 28891908
- [Derived] Hammond FM, Sherer M, Malec JF, Zafonte RD, Whitney M, Bell K, Dikmen S, Bogner J, Mysiw J, Pershad R; Amantadine Irritability Multisite Study Group. Amantadine Effect on Perceptions of Irritability after Traumatic Brain Injury: Results of the Amantadine Irritability Multisite Study. J Neurotrauma. 2015 Aug 15;32(16):1230-8. doi: 10.1089/neu.2014.3803. Epub 2015 Mar 31. PMID 25774566
- See also: Carolinas Rehabilitation — http://www.carolinasrehabilitation.org/
- See also: Carolinas HealthCare System — http://www.carolinashealthcare.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participant recruitment occurred 2009 - 2013 via referrals, letters from physicians, newsletters, and local brain injury support groups.
Period: Overall Study
Arm/Group | Amantadine | Placebo
Started | 82 | 86
Completed 28-day Mid-point | 80 | 81
Completed | 75 | 82
Not Completed | 7 | 4
Not completed — Lost to Follow-up | 2 | 1
Not completed — Withdrawal by Subject | 4 | 2
Not completed — Missed visit | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Amantadine | Placebo | Total
Number analyzed (Participants) | 82 | 86 | 168
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.18 (12.67) | 38.23 (12.36) | 39.21 (12.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 20 | 38
  Male | 64 | 66 | 130

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With >2-point Increase on Neuropsychiatric Inventory - Irritability Domain Rated by Observer Day 28
Description: The Neuropsychiatric Inventory (NPI) is a 40-item rating scale developed to assess 12 behavioral domains. Only the NPI-Irritability (NPI-I) domain was used for this study. NPI-I measures irritability with items including: bad temper, rapid mood changes, sudden anger, impatience, crankiness, argumentative. The rater selects the frequency (1-3) and severity (1-4) of the most problematic of these behavioral aspect(s) over the preceding month. The NPI score is the product of the frequency and severity for the NPI most problematic item score. The primary outcome measure was the proportion of participants with greater than two-point increase on the Neuropsychiatric Inventory Irritability domain. The total range is 1 (least irritability) - 12 (worst irritability).
Time Frame: Day 28
Measure: Number; unit: percentage of participants NPI improve>2
Arm/Group | Amantadine | Placebo
Number analyzed (Participants) | 80 | 81
percentage of participants NPI improve>2 | 66.3 | 66.7
Statistical Analysis 1: Comparison: Amantadine vs Placebo; Test type: Other; p = 0.9554, Chi-squared; Difference in percents = -0.4, 95% CI 2-sided [-14.7 to 13.9]

2. Secondary Outcome: Change in Neuropsychiatric Inventory - Irritability Domain Assessed by Observer Day 28
Description: as for outcome 1
Time Frame: Day 28
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Amantadine | Placebo
Number analyzed (Participants) | 80 | 81
score on a scale | -4 (3.39) | -4 (3.36)
Statistical Analysis 1: Comparison: Amantadine vs Placebo; Test type: Other; p = 0.96, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Proportion of Participants With >2-point Increase on Neuropsychiatric Inventory - Irritability Domain Rated by Participant Day 28
Description: as for outcome 1
Time Frame: Day 28
Measure: Number; unit: percentage of participants NPI improve>2
Arm/Group | Amantadine | Placebo
Number analyzed (Participants) | 80 | 81
percentage of participants NPI improve>2 | 51.3 | 40.5
Statistical Analysis 1: Comparison: Amantadine vs Placebo; Test type: Other; p = 0.1662, Chi-squared; Difference in percents = 10.8, 95% CI 2-sided [-4.2 to 25.8]

4. Secondary Outcome: Change in Neuropsychiatric Inventory - Irritability Domain Assessed by Participants Day 28
Description: as for outcome 1
Time Frame: Day 28
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Amantadine | Placebo
Number analyzed (Participants) | 80 | 81
score on a scale | -3 (3.58) | -2 (3.9)
Statistical Analysis 1: Comparison: Amantadine vs Placebo; Test type: Other; p = 0.3488, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Clinical Global Impressions Day 28
Description: Study physician's impression of change since study onset. Clinicians Global Impressions of Change (CGI) is a sensitive, standardized tool to assess psychopharmacologic treatment response completed by the study physician. The Global Improvement (GI) CGI subscale documented the clinician's impression of change. The GI uses a 7-point scale to assess beneficial and negative effects. Low GI values (1 -3) indicate improvement; higher values (4-7) represent worsening.
Time Frame: 28 Days
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Amantadine | Placebo
Number analyzed (Participants) | 80 | 81
score on a scale | 3.00 (1.14) | 3.00 (0.92)

6. Secondary Outcome: Proportion of Participants With >2-point Increase on Neuropsychiatric Inventory Irritability Domain Rated by Observers Day 60
Description: As described above for the primary measure, assessed as a secondary measure at Day 60. The Neuropsychiatric Inventory (NPI) is a 40-item rating scale developed to assess 12 behavioral domains. Only the NPI-Irritability (NPI-I) domain was used for this study. NPI-I measures irritability with items including: bad temper, rapid mood changes, sudden anger, impatience, crankiness, argumentative. The rater selects the frequency (1-3) and severity (1-4) of the most problematic of these behavioral aspect(s) over the preceding month. The NPI score is the product of the frequency and severity for the NPI most problematic item score. The primary outcome measure was the proportion of participants with greater than two-point increase on the Neuropsychiatric Inventory Irritability domain. The total range is 1 (least irritability) - 12 (worst irritability).
Time Frame: 60 days
Measure: Number; unit: percentage of participants NPI improve>2
Arm/Group | Amantadine | Placebo
Number analyzed (Participants) | 75 | 82
percentage of participants NPI improve>2 | 74.7 | 68.3
Statistical Analysis 1: Comparison: Amantadine vs Placebo; Test type: Other; p = 0.38, Chi-squared; Difference in percents = 6.4, 95% CI 2-sided [-7.2 to 20]

7. Secondary Outcome: Proportion of Participants With >2-point Increase on Neuropsychiatric Inventory - Irritability Domain Rated by Participant Day 60
Description: as for outcome 1
Time Frame: Day 60
Measure: Number; unit: percentage of participants NPI improve>2
Arm/Group | Amantadine | Placebo
Number analyzed (Participants) | 75 | 82
percentage of participants NPI improve>2 | 60.5 | 48.8
Statistical Analysis 1: Comparison: Amantadine vs Placebo; Test type: Other; p = 0.1373, Chi-squared; Difference in percents = 11.7, 95% CI 2-sided [-3.3 to 26.7]

8. Secondary Outcome: Change in Neuropsychiatric Inventory - Irritability Domain Assessed by Observers Day 60
Description: as for outcome 1
Time Frame: Day 60
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Amantadine | Placebo
Number analyzed (Participants) | 75 | 82
score on a scale | -5 (3.12) | -4 (3.42)
Statistical Analysis 1: Comparison: Amantadine vs Placebo; Test type: Other; p = 0.12, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Change in Neuropsychiatric Inventory - Irritability Domain Assessed by Participants Day 60
Description: as for outcome 1
Time Frame: Day 60
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Amantadine | Placebo
Number analyzed (Participants) | 75 | 82
score on a scale | -3 (2.83) | -2 (2.83)
Statistical Analysis 1: Comparison: Amantadine vs Placebo; Test type: Other; p = 0.0353, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Clinical Global Impressions Day 60
Description: as for outcome 5
Time Frame: 60 days
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Amantadine | Placebo
Number analyzed (Participants) | 82 | 75
score on a scale | 3.00 (1.05) | 3.00 (1.08)

ADVERSE EVENTS:
Arm/Group | Amantadine | Placebo
Serious Adverse Events (participants affected / at risk) | 3/82 | 2/86
Other Adverse Events (participants affected / at risk) | 36/82 | 33/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Amantadine (N=82) | Placebo (N=86)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Other infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Paranoia (Psychiatric disorders) | 1 (1) | 0 (0)
Other general medical (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Amantadine (N=82) | Placebo (N=86)
headache (Nervous system disorders) | 5 (5) | 2 (2)
Insomnia/ sleep disturbance (Nervous system disorders) | 7 (7) | 10 (10)
Connstipation (Gastrointestinal disorders) | 6 (6) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 5 (5) | 1 (1)
Other general medical (General disorders) | 10 (10) | 13 (13)
Other (General disorders) | 3 (3) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No